CLINICAL TRIAL: NCT04256044
Title: Analysis of Peripheral Blood ILC2s and Th2 Cells in Response to ANB020
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Medicines Evaluation Unit Ltd (Industry); AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0628
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Observational

SUMMARY:
This exploratory laboratory only study will assess alterations in immune cells in blood samples that may be responsive to an inflammatory mediator in asthma called IL-33 (Innate lymphoid type 2 cells, basophils and Th2 cells) in response to treatment with ANB020/placebo (a drug that targets IL-33, in the linked clinical trial ANB020-004). The study will involve additional 10ml blood draws on scheduled study visits in the ANB020-004 clinical trial at baseline, 1 week, 5 weeks, 18 weeks (4 visits total). Total number of subjects is 24 at the same 3 participating UK sites as the main linked clinical trial ANB020-004.

Blood samples will be sent on the same day to a flow cytometry laboratory at the NIHR Leicester Biomedical Research Centre (BRC) - Respiratory. A dedicated post doctoral, trained laboratory scientist will analyse the blood samples for the required cell types using a technique called flow cytometry - this technique identifies cell surface and intercellular markers, that together provide a unique cell identity. The experiments will be supervised by a senior research scientist and flow cytometrist Professor Dave Cousins, at the University of Leicester and results of the experiments will be fed back to AnaptysBio (the linked clinical trial Sponsor). Professor Salman Siddiqui at the University of Leicester will oversee the clinical conduct of this laboratory study and act as the Chief Investigator. Professor Siddiqui is also the local site lead Principal Investigator at Leicester for the linked ANB020-004 clinical trial described below.

The linked study (ANB020-004) is a Double-blind Placebo-Controlled Proof of Concept Study to Investigate ANB020 (a drug that targets an inflammatory mediator called IL-33) Activity in Adult Patients with Severe Eosinophilic Asthma. The expected duration of the study is up to 141 days. Screening period of 7-14 days and treatment and follow-up period of 127 days.

ELIGIBILITY:
Inclusion Criteria: Consenting participant in the ANB020-004 clinical trial (EudraCT 2017-000647-40) -

Exclusion Criteria:1) Unwilling to have four additional blood samples (10 mls per sample) for flow cytometry as part of the flow cytometry biomarker study linked to existing ANB020-004 study. (EudraCT 2017-000647-40)

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients taking part in the link study ANB202-004 (EudraCT 2017-000647-40) will be asked to take part in this observational study, in parallel with the main study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
To investigate whether treatment with ANB020, a drug that targets IL-33 alters levels of Basophils, Th2 cells or innate lymphoid type 2 cells (ILC2s) in peripheral blood | 18 weeks
  To investigate whether treatment with ANB020, a drug that targets IL-33 (an inflammatory mediator in asthma) alters levels of Basophils, Th2 cells or innate lymphoid type 2 cells (ILC2s) in peripheral blood in patients receiving active drug compared to placebo, in a linked clinical trial sponsored by AnaptysBio - ANB020-004.

CONTACTS AND LOCATIONS:
Overall Officials: David Cousins, Prof, Principal Investigator — University of Leicester
Locations (1):
- NIHR Leicester Biomedical Research Centre, Glenfield Hospital, Leicester, United Kingdom